CLINICAL TRIAL: NCT04341311
Title: Phase 1 Trial of Marizomib Alone and in Combination With Panobinostat for Children With Diffuse Intrinsic Pontine Glioma
Brief Title: Phase I Study of Marizomib + Panobinostat for Children With DIPG
Acronym: DIPG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawal of support from BMS
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Celgene (Industry); Secura Bio, Inc. (Industry)
Responsible Party: Principal Investigator, Katherine Warren, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-654
Record Dates: First submitted 2020-03-05; First posted 2020-04-10 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Pediatric Brainstem Glioma; Pediatric Brainstem Gliosarcoma, Recurrent; Pediatric Cancer; Pediatric Brain Tumor; Diffuse Glioma
Keywords: Diffuse Intrinsic Pontine Glioma; Pediatric Brainstem Glioma; Pediatric Cancer; Pediatric Brain Tumor; Diffuse Glioma; Progressive Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Recurrence; Neoplasms | interventions — marizomib; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Marizomib (Experimental): All patients will initially receive marizomib (MRZ) alone (Course A1) The dose escalation and de-escalation for single agent and combination will be guided using the Bayesian optimal interval (BOIN) design
  -Intravenously initially given every other week over a 28 day course but may go to weekly x 3 and weekly x 4 as the dose levels increase. Up to 26 courses.
  Interventions: Drug: Marizomib
- Marizomib + Panobinostat (Experimental): If tolerated,combination of Marizomib: and panobinostat on subsequent cycles. The dose escalation and de-escalation for single agent and combination will be guided using the Bayesian optimal interval (BOIN) design.
  * Intravenously initially given every other week over a 28 day course but may go to weekly x 3 and weekly x 4 as the dose levels increase. Up to 26 courses.
  * Panobinostat: Oral dosage is given 3 times weekly, every other week over a 28 day course
  Interventions: Drug: Marizomib; Drug: Panobinostat

INTERVENTIONS:
Drug: Marizomib — - Intravenously initially given every other week over a 28 day course but will go to weekly x 3 and weekly x 4 as the dose levels increase Up to 26 courses.
  Other Names: salinosporamide A; salinosporin A
Drug: Panobinostat — - Panobinostat: Oral dosage is given 3 times weekly, every other week over a 28 day course
  Other Names: Farydak
  Arms: Marizomib + Panobinostat

SUMMARY:
This research study is evaluating the safety, tolerability and preliminary efficacy of the drugs marizomib and panobinostat in pediatric patients with diffuse intrinsic pontine glioma (DIPG).

The names of the study drugs involved in this study are:

* Marizomib
* Panobinostat

DETAILED DESCRIPTION:
This research study involves chemotherapy as a possible treatment for pediatric patients with Diffuse intrinsic pontine glioma (DIPG)

* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
* The names of the study drugs involved in this study are:

  * Marizomib
  * Panobinostat

This study consists of 2 parts:

* Part A : The investigators are looking at the highest dose (up to a targeted maximum dose) of the study drug Marizomib that can be administered safely without severe or unmanageable side effects in participants that have DIPG, not everyone who participates in this research study will receive the same dose of the study intervention. The dose given will depend on the number of participants who have been enrolled prior and how well the dose was tolerated.
* Part B: Participants who tolerate Marizomib alone will be treated with Marizomib and panobinostat, but at lower dose of marizomib than the dose of marizomib when given alone.

Participants are expected to be on study treatment for up to 2 years followed for up to 5 years.

It is expected that up to 45 people will take part in this research study. This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

* Marizomib has not been approved by the U.S. Food and Drug Administration (FDA) as a treatment for any disease.

  -- This is the first time Marizomib will be given to children.
* Panobinostat has not approved by the U.S. Food and Drug Administration (FDA) for the treatment of diffuse intrinsic pontine glioma but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have DIPG, as defined below, to be eligible for this protocol. Given the poor prognosis of all patients with DIPG, patients may enroll at any point in their disease course provided they have received standard radiation therapy (also defined below) and meet all other eligibility requirements.
* DIPG is defined, for this study, as a diffusely infiltrative lesion with the epicenter in the pons, involving at least 2/3 of the pons as assessed by T2 or FLAIR imaging, and with no major or primary exophytic component, OR a pontine-based lesion that is biopsy proven non-pilocytic, WHO II-IV glioma. H3K27M status will be assessed in patients when tissue is available, but patients are eligible regardless of H3K27M status. (Biopsy will NOT be performed as part of this study).
* Standard radiation therapy is defined, for this study, as 54-60 Gy standard focal (photon or proton) radiation therapy, administered over 6 weeks (+/- 10 days). Patients who receive standard radiation therapy with concurrent chemotherapy may be eligible as long as other criteria are met.
* Patients must be < 22 years of age at the time of enrollment.
* Patient must be able to swallow capsules whole.
* Karnofsky Performance Scale (KPS, for ≥ 16 years of age) or Lansky Performance Scale (LPS, for < 16 years of age) assessed within 7 days prior to treatment initiation must be ≥ 50%. Patients who are unable to walk because of neurologic deficits, but who are up and awake in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have recovered (defined as < Grade 1 or baseline to meet otherwise defined eligibility criteria) from acute treatment-related toxicities of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Patients must have received their last fraction of radiation therapy at least 2 weeks prior to treatment initiation.
* Patients must have received their last dose of known myelosuppressive chemotherapy at least 21 days prior to enrollment (42 days if prior nitrosourea).
* Investigational/Biologic Agent/Immunotherapy (for agents that fit more than one category, i.e. biologic and immunotherapy, use the longest time-point indicated since last therapy to assess eligibility; contact PI or Study Chair if any questions):

  * Patient must have recovered (< Grade 1) from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment.

    * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur and discussed with the principal investigator.
  * Monoclonal antibody treatment and agents with known prolonged half-lives: At least three half-lives must have elapsed prior to enrollment due to the potential risk of pseudoprogression.
  * Checkpoint inhibitors, vaccine, or CAR T cell therapy: At least 3 months must have elapsed from last treatment prior to enrollment due to the risk of pseudo-progression.
  * Convection Enhanced Delivery (CED)

    * Patients must be at least 4 weeks from last CED procedure, have no permanent indwelling CED device, and no evidence of acute or ongoing intra-tumoral hemorrhage as demonstrated by gradient echo MRI. Additionally, patients must have recovered (< Grade 1) from any acute toxicity potentially related to the infused agent or procedure.
  * Intra-arterial therapy: Patient must be at least 4 weeks from most recent procedure, regardless of chemotherapeutic agent(s) infused and no evidence of acute or ongoing intratumoral hemorrhage as demonstrated by gradient echo MRI. Additionally, patients must have recovered (< Grade 1) from any acute toxicity potentially related to the infused agent or procedure.
  * Information regarding any prior investigational therapy or procedure, including (but not limited to) agent(s), dose, method of administration, dates of administration, concomitant therapies, all toxicities reported to date and anticipated toxicities, must be available for review by this study PI prior to patient enrollment. This includes any investigational therapy, including (but not limited to) those given in other countries or in private clinics.

If information on an investigational therapy is unavailable or the PI cannot assess ongoing potential risk of a prior therapy, the patient is not eligible.

* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,000/mm3
  * Platelets ≥ 100,000/ mm3 (unsupported, defined as no platelet transfusion within 7 days, and recovery from post-transfusion nadir)
  * Hemoglobin (Hgb) ≥ 8 g/dL (may receive transfusions)
  * Total bilirubin ≤ 2 times institutional upper limit of normal (ULN)
  * ALT(SGPT) < 3 x institutional upper limit of normal
  * Albumin ≥ 3 g/dL
  * Potassium within institutional normal range
  * Serum total calcium (correct for serum albumin) or ionized calcium within institutional normal range
  * Serum creatinine based on age/gender as noted in Table 2. Patients who do not meet the criteria in the table but who have a 24-hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m2 are eligible.

    * Table 2: Serum Creatinine for age/sex Serum Creatinine for age/sex Age Maximum Serum Creatinine (mg/dL) Male Female < 3 years < 0.8 < 0.8 3 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

      * 16 years 1.7 1.4 The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR(63) utilizing child length and stature data published by the CDC.
  * Left ventricular ejection fraction ≥ 50 by gated radionuclide study OR shortening fraction of ≥ 27% by echocardiogram
  * Patient must have a QTcF interval < 450 milliseconds (ms).
* Patients must be off all colony-forming growth factor(s) (i.e. filgrastim, sargramostim or erythropoietin) for at least 7 days prior to enrollment; 14 days must have elapsed if patients received PEG formulations.
* Patients must agree to avoid grapefruit or grapefruit juice and Seville (sour) oranges during the entire study as these are known to interfere with panobinostat pharmacokinetics.
* Pregnant and breastfeeding women are excluded from this study because marizomib and panobinostat's potential for teratogenic or abortifacient effects is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with marizomib or panobinostat, breastfeeding should be discontinued if the mother is treated with marizomib or panobinostat.
* The effects of marizomib and panobinostat on the developing human fetus are unknown. For this reason, women of child-bearing potential and men (including those who have had a vasectomy) must agree to use contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and up to 3 months for a female and 6 months for a male after the last dose of the drug (either marizomib or panobinostat, whichever is administered last). If you are able to become pregnant, you will have repeat pregnancy tests during the test. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have received > 60 Gy total radiation to the pons (e.g. patients who have received re-irradiation) due to potential increased risk of intratumoral hemorrhage
* Patients who have had prior bone marrow transplant or received marrow ablative therapy
* Patients with implanted CED catheters (e.g. Renshaw) due to inability to fully evaluate disease status
* Patients with a history of spinal radiation or those with an indication for acute spine radiation (e.g. significant cord compression) (Patients with leptomeningeal disease may be eligible but should be reviewed with study PI prior to enrollment).
* Patients with a history of disorientation, hallucinations or episodes of confusion (unless associated with a clear etiology, e.g. sedation, and fully resolved with no episodes in the 2 weeks prior to enrollment) since diagnosis of DIPG
* Patients with current or prior history of posterior reversible encephalopathy syndrome (PRES)
* Patients with significant (i.e. requiring active/ongoing treatment) GI dysfunction or GI disease, e.g. inflammatory bowel disease.
* Patients with chronic diarrhea or current diarrhea (≥ 4 stools/day).
* Patients with any clinically significant unrelated systemic illness (e.g. serious infections, mental illness, or significant cardiac, pulmonary, hepatic or other organ dysfunction), that, in the opinion of the investigator, would compromise the ability of the patient to tolerate protocol therapy or put them at additional risk for toxicity or would interfere with the study procedures, ability to assign attribution, or results.
* Any ventricular arrhythmias with the exception of benign premature ventricular contractions
* Patients known to be refractory to red blood cell or platelet transfusions. Patients who are receiving any other anticancer or investigational drug therapy
* Patients who are required to receive any medication listed in Appendix B or is otherwise known to significantly prolong the QTc interval. (Note: Loperamide use is acceptable at doses no higher than listed in this protocol).
* Patients who are taking cannabinoids, cannabinoid oils, any psychoactive supplement, narcotics, or any agent that can potentially cause hallucinations, disorientation, confusion or dizziness
* Patients/parents/caregivers must disclose all supplements and/or alternative therapies being administered to the patient. If unwilling or unable, patient is not eligible.
* Patients receiving enzyme-inducing antiepileptic drugs and/or valproic acid. Patients are eligible if they discontinue enzyme-inducing antiepileptic drugs and/or valproic acid prior to enrollment and have a washout period of least 5 half-lives.
* Patients who, in the opinion of the investigator, are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions
* Known or suspected hypersensitivity to marizomib or panobinostat
* Any patient who has the potential to receive a marizomib dose less than 0.2 mg

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) of marizomib as a single agent | 28 Days
  To determine the toxicity profile and any dose-limiting toxicity (DLT) of marizomib as a single agent at doses up to 0.8 mg/m2 , in children with DIPG
Dose-limiting toxicity (DLT) of marizomib in combination with panobinostat | 28 days
  To determine the toxicity profile and any DLT of marizomib at doses up to 0.8 mg/m2 when administered in combination with panobinostat to children with DIPG
Maximum Tolerated Dose of Marizomib (single agent) | 28 Days
  To estimate the maximum-tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of marizomib when administered as a single agent in children with DIPG
Maximum Tolerated Dose of Marizomib in combination with panobinostat | 28 Days
  To estimate the MTD or RP2D of marizomib when administered in combination with panobinostat in children with DIPG
Pharmacokinetic parameters-volume of the central compartment (Vc/F) | Day 1 Course A1
  Estimated using compartmental methods. Plasma drug concentrations and pharmacokinetic parameters will be presented in tabular and graphical form
Pharmacokinetic parameters-elimination rate constant (Ke), | Course A1, Day 1
  Estimated using compartmental methods. Plasma drug concentrations and pharmacokinetic parameters will be presented in tabular and graphical form
Pharmacokinetic parameters half-life (t1/2) | Course A1, Day 1
  Estimated using compartmental methods. Plasma drug concentrations and pharmacokinetic parameters will be presented in tabular and graphical form
Pharmacokinetic parameters-apparent clearance (CL/F) | Course A1, Day 1
  Estimated using compartmental methods Plasma drug concentrations and pharmacokinetic parameters will be presented in tabular and graphical form
Area under the plasma concentration time curve (AUC) | Course A1, Day 1
  Estimated using compartmental methods Plasma drug concentrations and pharmacokinetic parameters will be presented in tabular and graphical form

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS) | rPFS will be measured from the time of treatment initiation until the time of progressive disease or death from any cause in patients with an event up to 60 Months.
  Kaplan-Meier method
Overall survival (OS) | time from enrollment until death due to any cause up to 60 Months
  Kaplan-Meier method will be used to summarize the time-to-event endpoints, i.e. OS
Clinical Benefit Score | Baseline, Day 1 of every Cycle up to 2 years. One cycle is 28 days. Higher scores may indicate more clinical benefit.
  determined by combination of radiographic assessment, symptoms (patient/parent-reported), clinical (physician or NP) assessment, steroid use, ability to walk, and quality of life (QOL) measure

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Warren, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu